CLINICAL TRIAL: NCT01508247
Title: A Multiple-center Randomized Double-blind Placebo-controlled Phase 3 Clinical Trial to Assess the Efficacy and Safety of an Inactivated Vaccine (Vero Cell) Against EV71 in Chinese Children Aged 6-35 Months
Brief Title: A Clinical Trial to Assess the Efficacy and Safety of an Inactivated Vaccine (Vero Cell) Against EV71 in Chinese Children Aged 6-35 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Bejing Vigoo Biological Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT010
Record Dates: First submitted 2012-01-04; First posted 2012-01-11 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Hand, Foot and Mouth Disease; Herpangina; Other EV71-associated Diseases
Keywords: efficacy; safety; inactivated vaccine (Vero Cell) against EV71; EV71-associated diseases
MeSH Terms: conditions — Hand, Foot and Mouth Disease; Herpangina | interventions — Vaccines, Inactivated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vaccine against EV71 (Experimental): Inactivated vaccine (Vero Cell) against EV71 of 320U /0.5ml in 5000 children aged 6-35 months on day0, 28
  Interventions: Biological: inactivated vaccine (Vero Cell) against EV71
- placebo (Placebo Comparator): 0/0.5ml placebo in 5000 children aged 6-35 months on day0, 28
  Interventions: Biological: 0/0.5ml placebo

INTERVENTIONS:
Biological: inactivated vaccine (Vero Cell) against EV71 — inactivated vaccine (vero cell) against EV71, 320U /0.5ml, two doses, on day0, 28
  Arms: vaccine against EV71
Biological: 0/0.5ml placebo — 0/0.5ml placebo, two doses, on day0, 28
  Arms: placebo

SUMMARY:
Since its discovery in 1969, enterovirus 71 (EV71) has been recognised as a frequent cause of epidemics of hand-foot-mouth disease (HFMD) associated with severe neurological sequelae in a small proportion of cases. There has been a significant increase in EV71 epidemic activity throughout the Asia-Pacific region since 1997. Recent HFMD epidemics in this region have heen associated with a severe from of brainstem encephalitis associated with pulmonary oedema and high case-fatality rates.

The data from the phase 1 and 2 trials suggested that the inactivated EV71 vaccine had a clinically acceptable safety and good immunogenicity for healthy Chinese children and infants. According to the immunogenicity and safety results, the 320U with adjuvant with immunizing schedule of two doses (per 28 day) will be applied in phase 3 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Only subjects fulfilling all of the following criteria will be eligible for the study:

* Healthy children aged from 6 to 35 months old
* General good health as established by medical history and physical examination
* The subjects' guardians are able to understand and sign the informed consent
* Had never received the vaccine against EV71
* The subjects' guardians allow to comply with the requirements of the protocol
* Available for all visits scheduled in this study
* Subjects with temperature <=37.0°C on axillary setting

Exclusion Criteria:

Subjects will not be eligible for the study if any of the following criteria is met:

* Subject who has a medical history of HFMD
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Family history of seizures or progressive neurological disease
* Family history of congenital or hereditary immunodeficiency
* Severe malnutrition or hypogenesis
* Major congenital defects or serious chronic illness, including perinatal brain damage
* Autoimmune disease
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with IM injections or blood draws
* Asplenia, functional asplenia, or splenic excision
* History of asthma, angioneurotic edema, diabetes or malignant tumour
* History of thyroidectomy, or thyroid disease in last 12 months
* Any acute infections in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of other research vaccines or medicines in last 1 month
* Any prior administration of attenuated live vaccine in last 15 days
* Any prior administration of subunit or inactivated vaccines in last 7 days
* Under the anti-TB prevention or therapy
* Subjects with temperature >37.0°C on axillary setting
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Exclusion Criteria for the second dose:

Subjects will not be eligible for the second dose if any of following adverse events happened after the first dose. They can continue other process of the study without the second dose vaccination according to the opinion of the investigator.

* Had any serious adverse events related to the first dose of inactivated vaccine (vero cell) against EV71 within 7 days
* Hypersensitivity reactions after vaccination (including urticaria/rashes that occur within 30 minutes after inoculation)
* Anaphylaxis after vaccination
* Any confirmed or suspected autoimmune disease or immune deficiency diseases, including human immunodeficiency virus (HIV) infection
* Any condition that in the opinion of the investigator, or IRB

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10245 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
the incidence density of the EV71-associated diseases in the vaccine group and placebo group. | begin at day 56 up to 14 months
  compare the incidence density of the EV71-associated diseases between the vaccine group and placebo group in Chinese children aged 6-35 months.

SECONDARY OUTCOMES:
the frequency of all the adverse events in vaccine group and placebo group. | up to 14 months
  compare frequency of all the solicited events, unsolicited adverse events and serious adverse events between vaccine group and placebo group.
Seropositive rate of the vaccine group | 8 months after first vaccination
  calculate the seropositive rate of the vaccine group in Chinese children aged 6-35 months at month 8 after first vaccination.
Seroconversion rate of the vaccine group | 8 months after first vaccination
  calculate the seroconversion rate of the vaccine group in Chinese children aged 6-35 months at month 8 after first vaccination.
GMT of the vaccine group | 8 months after first vaccination
  calculate the geometric mean titre (GMT) of the vaccine group in Chinese children aged 6-35 months at month 8 after first vaccination.
Seropositive rate of the vaccine group | 14 months after first vaccination
  calculate the seropositive rate of the vaccine group in Chinese children aged 6-35 months at month 14 after first vaccination.
Seroconversion rate of the vaccine group | 14 months after first vaccination
  calculate the seroconversion rate of the vaccine group in Chinese children aged 6-35 months at month 14 after first vaccination.
GMT of the vaccine group | 14 months after first vaccination
  calculate the geometric mean titre (GMT) of the vaccine group in Chinese children aged 6-35 months at month 14 after first vaccination.
Seropositive rate of the vaccine group and placebo group | 28 days after the second vaccination
  compare the seropositive rate of the vaccine group and placebo group in healthy children aged 6-35 months.
Seroconversion rate of the vaccine group and placebo group | 28 days after the second vaccination
  compare the Seroconversion rate of the vaccine group and placebo group in healthy children aged 6-35 months.
GMT of the vaccine group and placebo group | 28 days after the second vaccination
  compare the geometric mean titre (GMT) of the vaccine group and placebo group in healthy children aged 6-35 months.
GMI of the vaccine group and placebo group | 28 days after the second vaccination
  compare the geometric mean fold increase (GMFI) of the vaccine group and placebo group in healthy children aged 6-35 months.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Cai Zhu, Master, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (4):
- China (4):
  - Donghai County Center for Disease Control and Prevention, Lianyungang, Jiangsu
  - Pizhou County-Level City Center for Disease Control and Prevention, Xuzhou, Jiangsu
  - Baoying County Center for Disease Control and Prevention, Yangzhou, Jiangsu
  - Chaoyang Distinct Center for Disease Control and Prevention, Beijing

REFERENCES:
- [Derived] Zhu W, Jin P, Li JX, Zhu FC, Liu P. Correlates of protection for inactivated enterovirus 71 vaccine: the analysis of immunological surrogate endpoints. Expert Rev Vaccines. 2017 Sep;16(9):945-949. doi: 10.1080/14760584.2017.1335603. Epub 2017 Jun 12. PMID 28548626
- [Derived] Wei M, Meng F, Wang S, Li J, Zhang Y, Mao Q, Hu Y, Liu P, Shi N, Tao H, Chu K, Wang Y, Liang Z, Li X, Zhu F. 2-Year Efficacy, Immunogenicity, and Safety of Vigoo Enterovirus 71 Vaccine in Healthy Chinese Children: A Randomized Open-Label Study. J Infect Dis. 2017 Jan 1;215(1):56-63. doi: 10.1093/infdis/jiw502. Epub 2016 Oct 17. PMID 28077584
- [Derived] Zhu FC, Meng FY, Li JX, Li XL, Mao QY, Tao H, Zhang YT, Yao X, Chu K, Chen QH, Hu YM, Wu X, Liu P, Zhu LY, Gao F, Jin H, Chen YJ, Dong YY, Liang YC, Shi NM, Ge HM, Liu L, Chen SG, Ai X, Zhang ZY, Ji YG, Luo FJ, Chen XQ, Zhang Y, Zhu LW, Liang ZL, Shen XL. Efficacy, safety, and immunology of an inactivated alum-adjuvant enterovirus 71 vaccine in children in China: a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2013 Jun 8;381(9882):2024-32. doi: 10.1016/S0140-6736(13)61049-1. Epub 2013 May 29. PMID 23726161